CLINICAL TRIAL: NCT01245881
Title: A Multicenter Study of Fractional Photothermolysis in the Treatment of Melasma
Brief Title: Fractional Photothermolysis for Treating Melasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laserklinik Karlsruhe (Other)
Collaborators: Laser and Skin Centre Potsdam, Potsdam, Germany (Unknown)
Responsible Party: Christian Raulin, MD, Laserklinik Karlsruhe, Karlsruhe, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LK-13-2010
Record Dates: First submitted 2010-11-19; First posted 2010-11-23 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Melasma
Keywords: controlled trial; fractional photothermolysis; laser surgery; melasma; pigment disorder
MeSH Terms: conditions — Melanosis; Pigmentation Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Treatment group (Experimental): Broad-spectrum UV block plus non-ablative 1,550-nm fractional treatment
  Interventions: Device: Non-ablative fractional photothermolysis laser
- Control group (Active Comparator)
  Interventions: Other: broad-spectrum sunblock (SPF 50+)

INTERVENTIONS:
Device: Non-ablative fractional photothermolysis laser — * Wavelength: 1,550 nm;
  * Energy: 15 mJ/MTZ;
  * Total coverage: 20%;
  * Total density: 1,048 MTZs/cm2;
  * Density per pass: 131 MTZ/cm2;
  * Number of passes: 8.
  Arms: Treatment group
Other: broad-spectrum sunblock (SPF 50+)
  Arms: Control group

SUMMARY:
In several observational studies, non-ablative fractional photothermolysis (FP) has been reported to bridge the gap between efficacy and tolerability in the treatment of melasma. While some beneficial effects have been attributed to non-ablative FP in treating melasma, methodological constraints (e.g., a limited number of patients; no control group assignment) impair efficacy assessment; currently published results neither allow researchers and clinicians to draw valid conclusions nor warrant recommendations for therapy. In particular, bias resulting from poorly designed trials may mislead clinicians into making a wrong decision and generate not only unnecessary treatment (i.e., costs), but also a risk of side effects for patients. Therefore, the purpose of this trial was to clarify the efficacy and safety of FP in the treatment of melasma as compared to the lone application of a sun-blocking lotion (SPF >50).

ELIGIBILITY:
Inclusion Criteria:

* Adults (female/male) with clinical evidence of melasma;
* Fitzpatrick skin phototype I-III;
* Ability and willingness to comply with the requirements of the protocol.

Exclusion Criteria:

* Pregnancy or nursing;
* Inability to avoid sun exposure for occupational reasons (e.g., gardeners);
* Known history or clinically relevant allergy to components of the sunscreen or topical anaesthetic;
* Use of topical retinoids within 3 months prior to study enrolment;
* Use of topical hydroquinone within 6 months prior to study enrolment;
* Use of topical corticosteroids within 1 month prior to study enrolment;
* Use of topical cosmetic depigmenting agents within 2 weeks prior to study enrolment;
* Laser surgery procedures within the treatment region during the last 12 weeks prior to enrolment;
* Coagulation disorders or anticoagulant treatment;
* Photo-sensitizing medication (e.g., tetracyclines, gold).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Melasma Area and Severity Index (MASI) at 12 weeks after final treatment | Pre-treatment and at final follow-up (12 weeks after last treatment session)

SECONDARY OUTCOMES:
Subjective assessment of treatment outcome (by patients) | Pre-treatment and at final follow-up
Patient satisfaction | Pre-treatment and at final follow-up
Side effects | At each follow-up visit (week 3, 6, 9, 12)

CONTACTS AND LOCATIONS:
Locations (1):
- Laserklinik Karlsruhe, Karlsruhe, Germany